CLINICAL TRIAL: NCT05602259
Title: PROspective Trial on EOsinophilia in Non-Small Cell Lung Cancer (NSCLC) (PROTEON).
Brief Title: PROspective Trial on EOsinophilia in Non-Small Cell Lung Cancer (NSCLC).
Acronym: PROTEON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Anne Sibille, Dr Anne Sibille, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/258
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eosinophil detection (Experimental): Eosinophils will be measured in blood, sputum, bronchoalveolar lavage if available and biopsies.
  Interventions: Diagnostic Test: induced sputum; Diagnostic Test: lung biopsy; Diagnostic Test: bronchoalveolar lavage; Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: induced sputum — After premedication with 400 μg inhaled salbutamol, sputum will be induced by inhalation of hypertonic (NaCl 3%) or isotonic (NaCl 0.9%) saline combined according to the FEV-1 value (> or ≤ than 65% predicted). Saline will be combined with additional salbutamol delivered by an ultrasonic nebulizer (Ultra-Neb 2000; Devilbiss, Somerset, PA, USA) with an output set at 0.9 ml/min. Each subject will inhale the aerosol for three consecutive periods of 5 min for a total of 15 min. For safety reasons, FEV-1 will be monitored throughout the induction and will be stopped if FEV-1 would fall by more than 20% from baseline.
Diagnostic Test: lung biopsy — As per standard practice, biopsies will be taken from the primary tumour site or from a metastatic site.
Diagnostic Test: bronchoalveolar lavage — When available, the remaining material from a patient's bronchoalveolar lavage will be collected.
Diagnostic Test: blood draw — As per standard practice, blood will be drawn from patients before and during treatment. Data on white blood cells will be collected.

SUMMARY:
This prospective study will examine eosinophils in various biological materials to compare the detection in those materials and ascertain the prognostic and predictive role of eosinophils in untreated non-small cell lung cancer patient.

ELIGIBILITY:
Inclusion Criteria:

* o All stages of NSCLC

  * Stage III-IV NSCLC eligible for ICI treatment
  * 18 years or older; non pregnant women
  * in stage III-IV: no previous ICI and before ICI (mono- or combination therapy) initiation
  * Signed informed consent
  * Clinical, biological and radiological evaluation at the CHU de Liège for at least 6 months following treatment initiation

Exclusion Criteria:

* Probable noncompliance with the follow-up requirements of the study (psychiatric condition, socio-economic factors)
* Inclusion in a clinical study contraindicating the enrolment in the PROTEON study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Detection of eosinophils in untreated non-small cell lung cancer patients | Baseline (pre-treatment)
  Concentration of eosinophils will be used in various bodily materials as described above.

SECONDARY OUTCOMES:
Prognostic and predictive value of eosinophils in non-small cell lung cancer patients | Baseline (pre-treatment) and, if immunotherapy, after 3 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No